CLINICAL TRIAL: NCT04474093
Title: Monolithic CAD/CAM Single Tooth Crowns Made From Different Ceramics: One Year Preliminary Results of a Randomized Clinical Trial
Brief Title: Monolithic CAD/CAM Single Tooth Ceramic Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Diler Deniz, Clinical Instructor, Prosthetic Dentistry, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA-16029; THD-2016-11741 (Other: ( Other Grant/Funding Number: HacettepeU Scientific Research Projects Coordination Unit ))
Record Dates: First submitted 2020-07-02; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Crowns (MeSH Unique ID: D003442), Single Tooth; Dental Porcelain (MeSH Unique ID: D003776)
Keywords: Zirconium-reinforced glass ceramics(ZRGC); Lithium disilicate glass ceramics(LGC); Resin infiltrated glass ceramics(RIGC); Monolithic single tooth restoration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zirconium-reinforced glass ceramics (ZRGC) (Active Comparator): 12 posterior single tooth crowns made from monolithic zirconium-reinforced glass ceramics(ZRGC). Restorations were evaluated prosthetic and periodontal criteria at baseline, after 6 and 12 months. While prosthetic evaluation was performed according to Modified US Public Health Service criteria; probing depth(PD), clinical attachment level(CAL), gingival bleeding time index(GBTI), gingival(GI) and periodontal index(PI) were used in periodontal evaluation.
  Interventions: Other: Zirconium-reinforced glass ceramics(ZRGC),Lithium disilicate glass ceramics(LGC), Resin infiltrated glass ceramics(RIGC)
- Lithium disilicate glass ceramics (LGC) (Active Comparator): Group 2: 12 posterior single tooth crowns made from monolithic lithium disilicate glass ceramics(LGC). Restorations were evaluated prosthetic and periodontal criteria at baseline, after 6 and 12 months. While prosthetic evaluation was performed according to Modified US Public Health Service criteria; probing depth(PD), clinical attachment level(CAL), gingival bleeding time index(GBTI), gingival(GI) and periodontal index(PI) were used in periodontal evaluation.
  Interventions: Other: Zirconium-reinforced glass ceramics(ZRGC),Lithium disilicate glass ceramics(LGC), Resin infiltrated glass ceramics(RIGC)
- Resin infiltrated glass ceramics (RIGC) (Active Comparator): 12 posterior single tooth crowns made from monolithic resin infiltrated glass ceramics(RIGC). Restorations were evaluated prosthetic and periodontal criteria at baseline, after 6 and 12 months. While prosthetic evaluation was performed according to Modified US Public Health Service criteria; probing depth(PD), clinical attachment level(CAL), gingival bleeding time index(GBTI), gingival(GI) and periodontal index(PI) were used in periodontal evaluation.
  Interventions: Other: Zirconium-reinforced glass ceramics(ZRGC),Lithium disilicate glass ceramics(LGC), Resin infiltrated glass ceramics(RIGC)

INTERVENTIONS:
Other: Zirconium-reinforced glass ceramics(ZRGC),Lithium disilicate glass ceramics(LGC), Resin infiltrated glass ceramics(RIGC)

SUMMARY:
With the development of Computer Aided Design and Computer Aided manufacturing (CAD / CAM) systems, all ceramic restorations have been used with high success rates during the past 30 years in order to eliminate the disadvantages of metal ceramic restorations. Based on these developments, in every passing days new ceramic materials has been added to dental market. The aim of the present study was evaluating clinical results of single-tooth ceramic crowns in the posterior region produced from three different monolithic ceramic materials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Individuals who have signed the informed consent form
* Periodontally stable patients
* Having devital teeth need to be restored in the posterior region
* Having natural dentition or minimally invasive restoration against the restored tooth.

Exclusion Criteria:

* Diagnosed patients with temporomandibular joint problems
* Insufficient supportive tooth tissue for restoration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Survival rate and success (changes over time) | 1 year (Baseline to 12 months)
  12 crowns were made from each group of three different ceramics: ZRGC, LDGC and RIGC. Thereafter, the restorations was evaluated in terms of any failure or loss of the restoration at any follow-up (6th and 12th months) periods. The results were obtained proportionally in percent (%).
Prosthetic evaluation changes | 1 year (Baseline to 12 months)
  As recorded at the baseline (0), each restoration was assessed according to the modified the United States Public Health Service (USPHS) Ryge Criteria for prosthetic evaluation by a calibrated prosthodontics.USPHS criteria is based on the following ratings: Color match (Alpha,Bravo, Charlie), cavosurface marginal discoloration (Alpha,Bravo, Charlie), secondary caries (Alpha,Bravo), anatomic contour (Alpha,Bravo, Charlie), marginal integrity (Alpha,Bravo, Charlie), surface texture (Alpha,Bravo, Charlie) and gross fracture (Alpha,Bravo, Charlie).
Periodontal evaluation changes | 1 year (Baseline to 12 months)
  Probing depth(PD): Probing depth is defined as the distance from the free gingival margin to the bottom of the periodontal pocket (mm).
  Clinical attachment level(CAL): The loss of CAL were measured and calculated by measuring recession and subtracting the periodontal probing depth (mm).
  Gingival bleeding time index(GBTI): The probe were swiped at apical portion of the gingival crevice from line angle interproximally and after 10 seconds assessed if there was bleeding or no bleeding on the mesial and distal (unit/tooth).
  Plaque index(PI, according to Silness and Löe, 1964): The total mean PI is the sum of the individual scores divided by the number of investigated sites. The thickness and extension of plaque were assessed (unit/tooth).
  Gingival index(GI, according to Löe, 1967): The total mean GI is the sum of the individual scores divided by the number of investigated sites. The GI for each tooth is the sum of the 4 individual scores divided by 4 (unit/tooth).

CONTACTS AND LOCATIONS:
Overall Officials: Diler DENİZ, DDS, MSD, Principal Investigator — Clinical Instructor; Güliz AKTAŞ, DDS,PhD, Study Director — Associate Professor; M.Barış GÜNCÜ, DDS,PhD, Study Chair — Associate Professor; Güliz N. GÜNCÜ, DDS,PhD, Study Chair — Professor

IPD SHARING:
Plan to Share IPD: No